CLINICAL TRIAL: NCT03659682
Title: Effect of GLPIR Stimulation on Neuroprotection and Inflammation in Parkinson's Disease
Brief Title: GLP1R in Parkinson's Disease
Acronym: GIPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Vidar Gundersen, Neurologist, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120262PARK
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Parkinson Disease
Keywords: GLP1R, neuroprotection, inflammation
MeSH Terms: conditions — Parkinson Disease; Inflammation | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: delayed start design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- semaglutide (Active Comparator): Ozempic- 1.0 mg administered subcutaneously once weekly
  Interventions: Drug: Semaglutide
- placebo (Placebo Comparator): Placebo, 1.0 mg administered subcutaneously once weekly
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — subcutaneous, 1.0 mg, weekly, 48 months

SUMMARY:
The purpose of the study is to test the neuroprotective and anti-inflammatory properties of semaglutide in idiopathic Parkinson's disease (PD)

DETAILED DESCRIPTION:
The trial is a single center, double-blind, placebo-controlled study. We plan to enroll 270 newly diagnosed patents with idiopathic Parkinson's disease (PD) over 2 years. The subjects that are enrolled in the study will be randomised to receive once a week self-administered subcutaneous injections of semaglutide (1.0 mg) or placebo in a 1:1 study design.

Semaglutide has been approved by the Food and Drug Administration (FDA) and European Medicines Agency to treat adults with type 2 diabetes. The treatment has not been approved for use in patients with PD. Semaglutide is a synthetic analogue of glucagon-like peptide 1 (GLP1), which stimulates GLP1 receptors (GLP1R). Stimulation of GLP1R in B-cells in the pancreas potentiates insulin secretion and contribute to blood glucose regulation. In the brain it is known that GLP1R stimulation in the hypothalamus contribute to appetite and body weight regulation. Besides these known GLP1R effects, GLP1R can inhibit production of pro-inflammatory cytokines in microglia, which in turn will stop/slow down degeneration of neurons in the brain. Another GLP1 agonist, exenatide, has been tested in patients with PD, showing significant improvement of motor symptoms. However, it could not be concluded whether this was caused by an symptomatic or neuroprotective effect.

Eligible participants will be treated with semaglutide or placebo for 24 months in a double blind period 1 of the study. Thereafter both groups will receive semaglutide for another 2 years in an open period 2 of the study. The study will measure effects of semaglutide on motor symptoms (assessed by changes in the MDS-UPDRS part III, and in levo-dopa equivalents), on nigrostriatal degeneration (assessed by changes in DAT-scan uptake), on cognitive function (assessed by MME and MOCA, on quality of life (assessed by EQFDQ, PDQ) and on non-motor symptoms of PD (assessed by NMSS).The tests will be performed at baseline, after 12, 24, 36 and 48 months of the study. Blood and cerebrospinal samples will be taken to analyse inflammatory markers, and to confirm penetration of semaglutide across the blood brain barrier.

ELIGIBILITY:
Inclusion Criteria:

We will include newly diagnosed patients with PD, age 40-75. Diagnosis of clinically established early PD will be made according to the new criteria set by the Movement Disorder Society (Berg D et al Mov Disord 2018). Enrolment must occur within a year from diagnosis. Before inclusion in the trial PD diagnosis must be supported by typical findings on dopamine transporter (DAT)scans.

Exclusion Criteria:

Patients will be excluded if they have chronic inflammatory brain disorders, as verified or diagnosed on brain magnetic resonance imaging (MRI). Cognitive impairment in PD will be excluded by way of Mini Mental Status (MMS, score < 25 points) and Montreal Cognitive Assessment (MOCA, score <25 points). The patients will be excluded if they have diabetes type 2 and cancer, especially if they or family members have familiar medullary thyroid carcinoma, or multiple endocrine neoplastic syndrome type 2 (MEN 2), as well as those having manifest kidney failure (see side effects below). The patients cannot receive long-term treatment with anti-inflammatory drugs, or other experimental drugs. Patients who are pregnant or breastfeeding are excluded.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-02 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor Function | 48 months
  MDS-UPDRS part 3 in OFF medication state

IPD SHARING:
Plan to Share IPD: Undecided